CLINICAL TRIAL: NCT03438968
Title: Women in Cardiac Rehabilitation: Optimizing the Training Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Vermont (Other)
Responsible Party: Principal Investigator, Philip Ades, Professor of Medicine, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 18-0008
Record Dates: First submitted 2018-02-13; First posted 2018-02-20 (Actual); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Exercise Training; Coronary Artery Disease; Women; Cardiac Rehabilitation
MeSH Terms: conditions — Coronary Artery Disease | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: At stress testing, cardiologist will not know group assignment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity aerobic training (Experimental): Individuals will exercise using a high-intensity interval exercise training protocol
  Interventions: Behavioral: Exercise training
- Standard Moderate continuous training (Active Comparator): Individuals will exercise using a standard moderate intensity continuous exercise training protocol
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Cardiac Rehabilitation exercise training

SUMMARY:
Cardiovascular disease (CVD) is highly prevalent in women resulting in 398,086 deaths annually. Even as women participate in traditional CR programs, data specificity and subsequent research have yet to emerge in a meaningful way so that women-centered CR can be better customized and their outcomes properly assessed. Aerobic fitness is a powerful predictor of prognosis in individuals with CVD yet there is evidence that women do not improve their peak VO2 as much as men during CR. We have designed a training program for women based upon past research with a goal of optimizing their training potential in CR. This program combines the utilization of a training technique termed high intensity interval training along with specific strength training exercises of the upper legs. We hypothesize that women, irrespective of age, would be capable of high intensity interval training to improve peak aerobic capacity in the CR setting. Furthermore, since women often have a deficit of thigh strength entering CR, and thigh strength correlates with endurance walking,strength training will also be included. The purpose of this study is to examine the value of high intensity interval training and strength training to maximize aerobic training response in CR for women. This may contribute to establishing specific protocols and training guidelines for future program design for women in CR. Since a set of comprehensive CR guidelines pertaining to women is lacking, it is hoped that the results of this study will help us develop exercise protocols and regimen to better structure and modulate CR programs for optimal benefit to women.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) is the foremost leading cause of death in women.1 More than 1 in 3 female adults are affected by CVD.2 Though the prevalence of CVD in women remains high, there is a relative paucity of research pertaining to women in Cardiac Rehabilitation (CR). Improvements in peak VO2 in CR are prognostically important 3-5 and several studies have shown that women increase their aerobic capacity in CR to a lesser degree than men.6,7 Even as women participate in many traditional CR programs, data specificity and subsequent research has yet to emerge in a meaningful way so that women-centered CR can be better customized and their outcomes properly assessed.

It is understood that women demonstrate a lower VO2 max than that of men8 on entry into CR which is often attributed to their smaller muscle mass, lower hemoglobin and blood volume, and smaller stroke volume relative to men.9 A finding of our previous study on aerobic capacity in patients entering cardiac rehabilitation revealed that values of peak VO2 on entry to CR were extremely low, particularly in women.6 It has been observed in the CR setting that women have lower physical function scores than men.10 Handgrip strength also differs between men and women.11 Baseline maximal exercise capacity of peak VO2 has been found to be the best predictors of baseline physical function score along with strength measures of leg press and bench press.10 Another study of ours revealed that while a peak VO2 below 15 was associated with high risk of annual all-cause mortality among men, a peak VO2 below 12 was associated with highest risk among women.12 Though women in another study had lower peak exercise capacities than men, they achieved similar relative improvements as a result of cardiac rehabilitation.13 Research in the field deserves further exploration as the results remain mixed. As women improve less than men in attaining peak VO2, we have put together a training program for women with a goal of optimizing their training potential in CR. This program combines the utilization of a training technique termed interval training along with specific strength training exercises of the legs. Previous studies that included both men and women with CAD have indicated that high intensity interval training might be more beneficial than moderate or standard intensity training in terms of improvements in aerobic fitness.14-16 However, the specificity of benefits for women remains rather elusive. Thus, studying variations in strength and power with appropriate interval training could help us attain better outcomes.

We hypothesize that women, irrespective of age, would be capable of high intensity interval training to improve peak aerobic capacity in the CR setting. Furthermore, since women often have a deficit of thigh strength entering CR, strength training will also be included. The purpose of this study is to examine the value of high intensity interval training and strength training to maximize aerobic fitness in Cardiac Rehabilitation for women. This may contribute to establishing specific protocols and training guidelines for future program design for women in CR. Since a set of comprehensive CR guidelines pertaining to women is lacking, it is hoped that the results of this study will help us develop exercise protocols and regimen to better structure and modulate CR programs for optimal benefit to women.

Study Design: Describe the research design, including a description of any new methodology and its advantage over existing methodologies.

This is a prospective study to be conducted at University of Vermont Cardiac Rehabilitation Center involving female cardiac patients. At entry to CR, data to be collected from patients participating in the study include: 1) Baseline characteristics such as age, body weight and height for calculation of BMI, systolic and diastolic blood pressure (rest), heart rate (rest, peak), medications, prior cardiac event etc., 2) Aerobic fitness assessment using a symptom-limited graded exercise tolerance test on treadmill to determine Peak metabolic equivalents (METs peak) and Peak VO2, 3) Strength measurement assessment using a single-repetition maximal lift (bench press for upper body and leg extension for lower body) and a handgrip dynamometer for handgrip strength, 4) Perceived exertion rate after each training session using BORG 6-20 scale18, 5) Self-reported physical functioning assessment using the Medical Outcomes Study Short Form-36 (MOS SF-36) survey questionnaire (0-100 scale) with 100 representing excellent physical functioning, 6) a co-morbidity score to determine the presence of peripheral vascular disease, cerebrovascular disease, chronic lung disease, or orthopedic limitations. If a co-morbid condition is present, it is quantified by severity as follows: 1, present but not exercising-limiting; 2, present and impacts on exercise performance; and 3, exercising-limiting; a total co-morbidity score ranging from 0 to 12 is to be determined for each participant, and 7) any "quality of life improvements" for participants as measured by the MacNew Heart Disease Health-Related Quality of Life Questionnaire.19 All of these measures with the exception of the MacNew questionnaire are collected on all CR entrants in the clinical setting.

The standard exercise training protocol will comprise of 3-one hour long sessions per week spanning 12 weeks, consisting of aerobic exercise and resistance training. Each session includes treadmill walking, rowing, cycling and aerobic exercise in the control group will be performed at an intensity of 70-85% of peak HR (moderate intensity) for a total of 45 minutes with rest periods as needed between equipment Patients will also participate in resistance training which will include 1 set of 10 repetitions at an intensity of 60-65% of the single repetition maximal lift (1-RM) of the following: leg extension, leg curl, bench press, shoulder press, lateral pull down, and bicep curl. For those who underwent CABG, upper body resistance training will take place 3 months post-operatively.

The high intensity interval training with more intensive strength training will consist of 3-one hour sessions over the course of 12 weeks. For this group, all aerobic training will comprise of "high intensity interval treadmill walking" (HIT). Patients will warm up for 5 minutes at 60-70% of peak HR followed by 4 minute intervals to achieve 90-95% of peak HR. In between each interval will be a 4 minute walking period at 50-60% of peak HR. You will also perform other types of exercise such as cycling and rowing for up to a total of 45 minutes of aerobic exercise. You can rest, as needed, in between different types of exercise equipment. Additionally, this group will undergo strength training as described above, however, they will do 2 sets of 10 repetitions for upper leg exercises at an intensity of 80% 1-RM.

At entry to CR, the study participants will be asked to fill out the following questionnaires:

1. Medical Outcomes Study Short Form-36 (MOS SF-36) survey questionnaire to report the physical functioning
2. MacNew Heart Disease Health-Related Quality of Life Questionnaire to measure quality of life improvement

At the completion of the study after 12 weeks, the participants will be asked to do the same measures. Random IDs will be given to patients filling out the survey instruments to maintain privacy and confidentiality. Additionally, the results will be stored on a password-protected secure computer network of UVMMC.

Statistical Considerations:

Power calculations undertaken by us (80% power with 5% level of significance) based on Wisloff study15 suggested that a sample size of 19 per group is needed to detect a difference of 30% between groups in Peak VO2 by exercise training regimen. We intend to conduct an interim updated power analysis once we have 10 patients to better fine tune the power analysis.

Baseline characteristics will be presented as mean SD. Non- paired t-tests will be used for comparison between groups at baseline (pre-test), at the conclusion of the study (post-test), and percent changes after exercise regimen. ANOVA for repeated measures will be used for analyzing the effect of the exercise regimen between groups. A level of significance of P<0.05 will be used to indicate statistical significance.

All eligible participants in the study will perform the CR exercise training under the supervision of exercised physiologists. This study presents minimal risk to participants as indeed, CR participation yields a 25% decrease in overall mortality and a 31% decrease in hospitalizations in year 1.20

Benefits of CR include improved overall cardiovascular health, knowledge of physical functioning opportunities and limitations, and ability to both undertake and continue exercise for a longer span of time beyond the end of the study. An underlying assumption of the study is optimization of exercise might yield a greater training increase in Peak VO2 in the HIT group along with possible greater improvements in fitness and quality of life.

Both groups will obtain all of the standard benefits of CR which include a lower mortality rate, a lower re-hospitalization rate, and an improved quality of life.

Data Safety and Monitoring:

Hard copy of paper data will be stored in locked office and file cabinets. All electronic data will be password protected and stored on the UVMMC secured network server.

ELIGIBILITY:
Inclusion Criteria: Heart disease, eligible for cardiac rehabilitation -

Exclusion Criteria: Peak VO2 < 12 ml/kg/min

-

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Estimated)
Dates: Start 2017-08-24 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
Aerobic Fitness | 4-month study participation
  Peak VO2 measured with cardiopulmonary exercise testing

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont College of Medicine, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Khadanga S, Savage PD, Pecha A, Rengo J, Ades PA. Optimizing Training Response for Women in Cardiac Rehabilitation: A Randomized Clinical Trial. JAMA Cardiol. 2022 Feb 1;7(2):215-218. doi: 10.1001/jamacardio.2021.4822. PMID 34817540